CLINICAL TRIAL: NCT02475304
Title: A Randomized, Double Blind, Placebo-controlled Proof-of-concept Study of FP187 in Patients With Mild to Moderate Psoriatic Arthritis
Brief Title: Proof-of-concept Study of Forward Pharma (FP)187 in Patients With Mild/Moderate Psoriatic Arthritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficulties to enrol patients
Sponsor: Skane University Hospital (Other)
Responsible Party: Principal Investigator, Elke Theander, senior consultant Rheumatology, associate professor, PhD, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSA-201-DMF
Record Dates: First submitted 2015-05-31; First posted 2015-06-18 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Dimethyl Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental FP187 (Experimental): Treatment with a daily dose of 500mg FP187 (twice daily). Other names: Dimethyl fumarate
  Interventions: Drug: FP187
- Placebo Comparator (Placebo Comparator): Patients will receive the same number of tablets as patients randomized to FP187 arm in order to maintain the blind. The colour and shape of the FP187 and placebo tablets will be the same so that no visible difference is detectable
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FP187 — FP 187 is given as oral tablets twice daily, 500 mg daily
  Other Names: Dimethyl Fumarate
  Arms: Experimental FP187
Drug: Placebo
  Arms: Placebo Comparator

SUMMARY:
The purpose of this study is to investigate, whether FP187 is effective in the treatment of mild to moderate psoriatic arthritis.

DETAILED DESCRIPTION:
The study is randomised, double blind, placebo-controlled proof-of-concept trial to investigate the efficacy and safety of FP187 compared to placebo over 24 weeks of treatment in patients with mild to moderate psoriatic arthritis (PsA). The daily dose levels in the FP187 arm will be 500 mg. After completion of the double blind treatment of 24 weeks, all patients irrespective of their treatment arm will be switched to an additional 24 week open-label treatment phase with 500 mg / day FP187. Patient who do not complete the 24 week double blind part of the study as scheduled will not be eligible for participation in the open-label part.

ELIGIBILITY:
Inclusion Criteria:

* documented clinical diagnosis of mild to moderate psoriatic arthritis of at least 3 months
* active psoriatic arthritis with at least 2 tender and 2 swollen joints
* signed informed consent
* willingness and ability to comply with study procedures
* besides psoriatic arthritis, patient must be in good general health in the opinion of the investigator, as determined by medical history, physical examination, vital signs, electrocardiography and clinical laboratory parameters
* if patients are using methotrexate, they should be on a stable dosis of not more the 20mg per week for at least 90 days prior to study entrance and should present no serious toxic side effects attributable to methotrexate
* female of childbearing age must be either surgically sterile or use a highly effective medically accepted contraceptive method

Exclusion Criteria:

* female patients who are pregnant of breast-feeding or planning to become pregnant during the entire trial period
* male patients planning pregnancy with their partner during the entire trial period, or practicing unprotected sexual relationship during the entire trial period
* known allergy to any of the constituents of the products being tested
* known immunosuppressive diseases (e.g. HIV, AIDS)
* known history of latent or active granulomatous infection including tuberculosis, histoplasmosis or coccidioidomycosis
* presence of another inflammatory disease including but not limited to rheumatoid arthritis, ankylosing spondylitis, systemic lupus erythematous or Lyme disease
* presence of chronic widespread pain syndrome
* patients with pustular forms of psoriasis, erythrodermic or guttate psoriasis
* patients with another non-psoriatic arthropathy (e.g. osteoarthritis)
* presence of another serious or progressive disease including skin malignancy
* presence or history of any malignancy (except for basal cell carcinoma, squamous cell carcinoma in situ of the skin treated with no evidence of recurrence within 5 years, or cervix cancer in situ treated with no evidence of recurrence.)
* use at any time of an biological Disease Modifying Antirheumatic Drug (bDMARD) such as etanercept, adalimumab, golimumab, certolizumab pegol or infliximab
* corticosteroid injections within 12 weeks
* use of any dimethyl fumarate (DMF) containing product within 12 weeks
* use of any retinoid treatments, other immunosuppressive treatments, cytostatics or drugs with known harmful effects on the kidneys within the last 3 months
* use of cyclosporine, corticosteroids or psoralen + UVA (PUVA) treatment within 4 weeks
* ongoing stomach or intestinal problems (e.g. gastritis or peptic ulcer)
* Aspartate transaminase (AST) or Alanine transaminase (ALT) > 2x upper normal normal limit (UNL) or Gamma Glutamyl Transferase (gamma-GT) results >2.5 UNL
* estimated creatinine clearance (Cockcroft-Gault) < 60ml/min
* leucopenia (leucocyte count < 3.5/nl), eosinophilia (>750 / micro l) or lymphocytopenia (<1.02 / nl)
* protein detected by urine stick test
* participation in another clinical trial during the last 2 months or participation in a trial with another psoriatic arthritis treatment within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-05; Primary Completion 2016-10 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
American Congress of Rheumatology (ACR)20 | Week 24
  Proportion of patients with a 20% improvement from baseline in tender/swollen joint counts according to the American College of Rheumatology criteria (ACR) based on a 66/68 joint count.

SECONDARY OUTCOMES:
ACR 20 | Weeks 8, 12, 28, 36, 40, 52
  Proportion of patients with a 20% improvement from baseline in tender/swollen joint counts according to the American College of Rheumatology criteria (ACR) based on a 66/68 joint count.
BSA | Weeks 8, 12, 24, 28, 36, 40, 52
  Body Surface Area (BSA) affected by psoriasis
LEI | Weeks 8, 12, 24, 28, 36, 40, 52
  Change from baseline in the Leeds Enthesitis Index (LEI)
ACR 50 | Weeks 8, 12, 24, 28, 36, 40, 52
  Proportion of patients with a 50% improvement from baseline in tender/swollen joint counts according to the American College of Rheumatology criteria (ACR) based on a 66/68 joint count.
ACR 70 | Weeks 8, 12, 24, 28, 36, 40, 52
  Proportion of patients with a 70% improvement from baseline in tender/swollen joint counts according to the American College of Rheumatology criteria (ACR) based on a 66/68 joint count.
Pain | Weeks 8, 12, 24, 28, 36, 40, 52
  Change from baseline in Pain Visual Analogue Scale (VAS) score
EQ-5D | Weeks 8, 12, 24, 28, 36, 40, 52
  Change from baseline in European Quality of Life - 5 Dimensions (EQ-5D) score
BASDAI | Weeks 8, 12, 24, 28, 36, 40, 52
  Change from baseline in Bath Ankylosing Spondylitis Disease Activity (BASDAI) score
BASFI | Weeks 8, 12, 24, 28, 36, 40, 52
  Change from baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) score
HAQ | Weeks 8, 12, 24, 28, 36, 40, 52
  Change from baseline in Health Assessment Questionnaire (HAQ) score

CONTACTS AND LOCATIONS:
Overall Officials: Elke Theander, MD. PhD, Principal Investigator — Skåne University Hospital, Lund University, 20502 Malmö, Sweden
Locations (1):
- Department of Rheumatology, Skåne University Hospital, Malmo, Sweden